CLINICAL TRIAL: NCT00002293
Title: Nystatin Pastille for the Prophylaxis of Oral Candidiasis in Patients With AIDS or AIDS Related Syndromes
Brief Title: A Study of Nystatin in the Prevention of Fungal Infections of the Mouth in Patients With AIDS or AIDS-Related Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: 026B; 5
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: Nystatin; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Candidiasis, Oral
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nystatin

INTERVENTIONS:
Drug: Nystatin

SUMMARY:
To determine a safe, effective, and convenient dosing schedule for nystatin pastilles in the prophylaxis of oral candidiasis in patients with AIDS or AIDS related syndromes (group III or IV, CDC classification)

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Experimental drugs (IND drugs) which are targeted specifically against the AIDS virus or which stimulate the immune system.
* Systemic or oral antibiotics.

Patients must have AIDS or AIDS-related syndromes (HIV infection:

* Group III or IV, CDC classification) and not have been treated for oral candidiasis during the past year.
* Patients can be entered into the study who have:
* Other oral lesions due to Kaposi's sarcoma, herpes zoster, and herpes simplex.
* A positive or negative oral culture for Candida.
* Must be able to follow instructions regarding the use of a pastille.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Oral lesions diagnostic of oral candidiasis or systemic candidiasis.
* Suspected or proven candidal esophagitis.

Patients with the following are excluded:

* Oral lesions diagnostic of oral candidiasis or systemic candidiasis.
* Receiving any effective antifungal agent orally or intravenously within 72 hours of study entry.
* Not expected to survive for at least 6 months.
* Unable to voluntarily maintain a pastille in the buccal cavity for approximately 20 minutes twice a day.
* Known hypersensitivity to nystatin.
* Suspected or proven candidal esophagitis.

Prior Medication:

Excluded within 72 hours of study entry:

* Any oral or intravenous antifungal agent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Birmingham Veterans Administration Med Ctr / Univ of Alabama, Birmingham, Alabama
  - Bristol - Myers Squibb Co, Princeton, New Jersey

REFERENCES:
- [Background] MacPhail LA, Hilton JF, Dodd CL, Greenspan D. Prophylaxis with nystatin pastilles for HIV-associated oral candidiasis. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Aug 15;12(5):470-6. doi: 10.1097/00042560-199608150-00005. PMID 8757423